CLINICAL TRIAL: NCT06891235
Title: Oral Fluid Testing to Assess Cannabis Non-Use in Remote Clinical Trials
Brief Title: Study of Oral Fluid Testing Approach
Acronym: SOFTA
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lydia Shrier, Research Director, Boston Children's Hospital
Other Study IDs: IRB-P00050265
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cannabis Use; Cannabis Intoxication; Cannabis Use Disorder
Keywords: cannabis use; young adult; oral fluid testing
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective community sample: Community sample of 200 younger adults aged 18-30 years who have used cannabis in the past 30 days, report use frequency of ≥1x/week, and have a positive test for urinary 11-nor-9-carboxy-delta-9-tetrocannabinol (THC-COOH) at baseline
  Interventions: Other: Biologic testing for THC

INTERVENTIONS:
Other: Biologic testing for THC — Participants will be asked to complete at-home urine test(s) and a series of oral fluid tests.

SUMMARY:
The purpose of this study is to identify and evaluate oral fluid testing as a biologic measure of cannabis use days that can be assessed remotely. The researchers will conduct this fully virtual study among a community sample of 200 individuals aged 18-30 years who have used cannabis at least 1 time per week on average in the past 30 days. Participants will complete oral fluid (saliva) tests, urine tests, and Timeline Follow-back interviews (self-report) that indicate their recent cannabis use (delta-9-THC). Participants will present for 3 virtual study visits and be asked to complete activities in between: Study Visit 1 (Day 0; informed consent, baseline survey, TLFB interview), Study Visit 2 (~Day 3; TLFB interview, urine testing), 6 days of at-home videorecorded oral fluid testing, Study Visit 3 (~Day 12; TLFB interview, urine test, oral fluid test, survey, interview).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30 years
* Cannabis use on >=1x/week in the past 30 days
* Ownership of a portable device that is capable of videoconference and videorecording (i.e., smartphone, tablet computer, or laptop computer)
* Ability to read and speak English
* Availability for duration of the study (2-3 weeks).
* To proceed to oral fluid testing, positive result for urinary TCH-COOH

Exclusion Criteria:

• Inability/unwillingness to provide contact information

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Testing duration: self-testing | Across 6 days leading up to the Day-12 visit
  Duration in minutes of videos of self-testing
Testing duration: observed test | Day of/During the Day-12 visit
  Duration in minutes of observed self-testing during study visit
Oral fluid testing protocol adherence: self-testing completed | Across 6 days leading up to the Day-12 visit
  Number and percent of videos of self-testing completed
Oral fluid testing protocol adherence: observed test completed | Day of/During the Day-12 visit
  Number and percent of live self-testing completed
Oral fluid testing protocol adherence: testing steps performed | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Number and percent of each step of self-testing performed (yes/no)
Oral fluid testing protocol adherence: testing steps performed correctly | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Number and percent of each step of self-testing performed correctly (yes/no)
Unreadable test results | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Number and percent of oral fluid tests with unreadable results
Inconclusive test results | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Number and percent of oral fluid tests with inconclusive results
Oral fluid test results | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Oral fluid test results for delta-9- tetrahydrocannabinol (delta-9-THC) on day of test (negative = non-use / positive = use)
Oral fluid acceptability | Day-12 visit
  Measure of acceptability (usability, likability, burden), 5 items, 5-point Likert-type scale (1, Strongly Disagree to 5, Strongly Agree), with higher score indicating greater acceptability.
  Benchmark for scale: ≥80% of participants with mean item score ≥4 out of 5
Use/Non-use intervals of 4 days | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Agreement between oral fluid results for 3 consecutive days (any positive = use / all negative = non-use) and self-report on timeline follow-back (TLFB) calendar interview for the same 3 days plus 1 day earlier (any days of use = use / no days of use = non-use).
  Benchmark: ≥ moderate agreement (Cohen's kappa ≥ 0.6)
Use/Non-use | Day-12 visit
  Agreement between oral fluid test results (positive/negative) and urine test result (positive/negative).
  Benchmarks: strong agreement (Cohen's kappa ≥ 0.8) for use; weak agreement (Cohen's kappa < 0.6) for non-use

SECONDARY OUTCOMES:
Use/Non-use for intervals of 2-8 days | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Agreement (use/non-use) between oral fluid test results and cannabis use reported on TLFB calendar interview for corresponding intervals ranging from 2 days (day of and day before testing, ≤24 hours prior) to 8 days

OTHER OUTCOMES:
Within-day frequency of cannabis use | Day-12 visit
  Number of times cannabis used within each day included in the intervals being examined for agreement (Specific Aim 2A and 2B), reported on TLFB calendar interview
Timing of cannabis use | Across 6 days leading up to the Day-12 visit; Day of/During the Day-12 visit
  Number of hours between last use and oral fluid testing time

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified survey data and biologic test result data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified scientific data will be shared as soon as possible. De-identified scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: De-identified scientific data and metadata arising from the project will be archived in the openICPSR repository. De-identified scientific data from this project will be findable through summary information (metadata) that will be readily available on the Center for Adolescent Behavioral Health Research website, the repository website, and clinicaltrials.gov.